CLINICAL TRIAL: NCT04961645
Title: Brain Stimulation Study of Human Visually-guided Navigation Using Repetitive Transcranial Magnetic Stimulation (rTMS)
Brief Title: Brain Stimulation and Visually-guided Navigation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated in February 2025 after interim analyses among participants in the computer-based task study arm showed that the rTMS was not a successful method of evaluating involvement of OPA in visually-guided navigation.
Sponsor: Emory University (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Daniel Dilks, Associate Professor, Emory University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00002512; 5R01EY029724 (NIH)
Record Dates: First submitted 2021-07-05; First posted 2021-07-14 (Actual); Results first posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Healthy Participants
Keywords: Visually-guided navigation
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: The computer-based task study arm will occur first prior to enrolling participants into the behavioral-based task study arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Repetitive Transcranial Magnetic Stimulation (rTMS) During Computer-based Task (Experimental): Participants receiving rTMS while they perform computer-based tests to examine the causal involvement of OPA in visually-guided navigation. The study visit lasts approximately 90 minutes.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS); Behavioral: Computer-based Test
- Repetitive Transcranial Magnetic Stimulation (rTMS) During Behavioral-based Task (Experimental): Participants receiving rTMS while they perform behavioral-based tests to examine the causal involvement of OPA in visually-guided navigation. The study visit lasts approximately 90 minutes.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS); Behavioral: Behavioral-based Test

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — TMS is a safe and noninvasive method for affecting brain function relying on the properties of electromagnetic induction. Action potentials are triggered in neurons, along with a subsequent period of deactivation. Normal ongoing brain activity is disrupted providing a way for investigators to produce a transient and reversible period of brain disruption.
Behavioral: Computer-based Test — Participants will be seated comfortably in a chair and asked to complete a simple computer-based task where they imagine walking through a room and press a button indicating if they can leave through a door on the left, center, or right wall. During or just before each of these tasks, participants will receive rTMS. In rTMS, a small plastic coil is placed next to the participant's head. The coil will be placed over the relevant brain region identified during the participant's fMRI scan. The coil will then generate a magnetic pulse, and stimulation will occur.
  Arms: Repetitive Transcranial Magnetic Stimulation (rTMS) During Computer-based Task
Behavioral: Behavioral-based Test — Participants will be asked to complete a simple behavioral task that will require them to walk around in a small room and search for hidden objects. During or just before each of these tasks, participants will receive rTMS. In rTMS, a small plastic coil is placed next to the participant's head. The coil will be placed over the relevant brain region identified during the participant's fMRI scan. The coil will then generate a magnetic pulse, and stimulation will occur.
  Arms: Repetitive Transcranial Magnetic Stimulation (rTMS) During Behavioral-based Task

SUMMARY:
This study investigates the neural mechanisms causally involved in how people navigate through their immediately visible environment (e.g., walking around one's bedroom flawlessly and effortlessly, not bumping into the walls or furniture). To investigate whether particular neural mechanisms are causally involved in "visually-guided navigation", repetitive transcranial magnetic stimulation (rTMS) is used to temporarily disrupt the functioning of particular brain regions in healthy adults while they are shown simple visual stimuli of places (e.g., bedrooms, kitchens, and living rooms) and asked to perform simple computer tasks or to complete simple behavioral tasks.

DETAILED DESCRIPTION:
Human ability to navigate through the immediately visible environment is crucial for survival. However, the representations and computations underlying this remarkable ability are not well understood, and current computer vision algorithms (robots) still lag far behind human performance. One promising strategy for attempting to understand "visually-guided navigation" is to characterize the neural systems that accomplish it. The results from functional magnetic resonance (fMRI) on adult humans have begun to elucidate the cortical regions involved in visually-guided navigation, with the central finding that there is at least one visual cortical region - called the occipital place area (OPA) that may play a central role in the ability to navigate through currently visible places (e.g., walking around our bedroom flawlessly and effortlessly, not bumping into the walls or furniture our bedroom). However, fMRI is a correlational method, and research still needs to determine if this functionally specific brain region is causally involved in visually-guided navigation. Understanding the causal involvement of this region will provide important clues about how humans navigate their world, and also perhaps someday be harnessed to help those individuals who devastatingly lose the ability to navigate, as a result of eye diseases, brain surgery, stroke, neurodegenerative diseases, or developmental disorders.

The use of rTMS to investigate the causal involvement of particular brain regions in particular human abilities is not novel, having been used to investigate face recognition, scene recognition, and object recognition. The general question for this research is to determine, using rTMS, the causal involvement of OPA in visually-guided navigation.

Participants will have an fMRI scan to identify the OPA location in each individual participant. Once the OPA location is known, participants will receive the rTMS study intervention.

ELIGIBILITY:
Inclusion Criteria:

* Normal or corrected-to-normal vision

Exclusion Criteria:

* Metal in the body
* Personal or first-degree family history of epileptic seizure
* A known brain injury
* Claustrophobia
* Taking certain medications that may increase the risk of seizures (e.g., bupropion, varenicline, chlorpromazine, theophylline) or reduce the effects of rTMS, such as benzodiazepines
* Adults who are unable to consent, pregnant women, and prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2023-03-03 (Actual); Primary Completion 2023-05-17 (Actual); Study Completion 2023-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Dilks, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at Emory University in Atlanta, Georgia, USA. Participant enrollment began March 3, 2023 and the final study visit occurred May 17, 2023. The study was terminated in February 2025. The study was terminated prior to enrolling participants into the behavioral-based task study arm.
Groups:
- Repetitive Transcranial Magnetic Stimulation (rTMS) During Computer-based Task: Participants receiving rTMS while they perform computer-based tests to examine the causal involvement of OPA in visually-guided navigation. The study visit lasts approximately 90 minutes.
  Repetitive Transcranial Magnetic Stimulation (rTMS): TMS is a safe and noninvasive method for affecting brain function relying on the properties of electromagnetic induction. Action potentials are triggered in neurons, along with a subsequent period of deactivation. Normal ongoing brain activity is disrupted providing a way for investigators to produce a transient and reversible period of brain disruption.
  Participants will be seated comfortably in a chair and asked to complete a simple computer-based task. During or just before each of these tasks, participants will receive rTMS. In rTMS, a small plastic coil is placed next to the participant's head. The coil will be placed over the relevant brain region identified during the participant's functional magnetic resonance (fMRI) scan. The coil will then generate a magnetic pulse, and stimulation will occur.
- Repetitive Transcranial Magnetic Stimulation (rTMS) During Behavioral-based Task: Participants receiving rTMS while they perform behavioral-based tests to examine the causal involvement of OPA in visually-guided navigation. The study visit lasts approximately 90 minutes.
  Repetitive Transcranial Magnetic Stimulation (rTMS): TMS is a safe and noninvasive method for affecting brain function relying on the properties of electromagnetic induction. Action potentials are triggered in neurons, along with a subsequent period of deactivation. Normal ongoing brain activity is disrupted providing a way for investigators to produce a transient and reversible period of brain disruption.
  Participants will be seated comfortably in a chair and asked to complete a simple behavioral task that will require them to walk around in a small room. During or just before each of these tasks, participants will receive rTMS. In rTMS, a small plastic coil is placed next to the participant's head. The coil will be placed over the relevant brain region identified during the participant's fMRI scan. The coil will then generate a magnetic pulse, and stimulation will occur.
Period: Overall Study
Arm/Group | Repetitive Transcranial Magnetic Stimulation (rTMS) During Computer-based Task | Repetitive Transcranial Magnetic Stimulation (rTMS) During Behavioral-based Task
Started | 11 | 0
Completed | 11 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Repetitive Transcranial Magnetic Stimulation (rTMS) During Computer-based Task: Participants receiving rTMS while they perform computer-based tests to examine the causal involvement of OPA in visually-guided navigation.
Arm/Group | Repetitive Transcranial Magnetic Stimulation (rTMS) During Computer-based Task
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 2
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Accuracy During Visually-guided Navigation Computer-based Task
Description: To assess performance during the visually-guided navigation computer-based task, rTMS is applied to to the control vertex site, which is not implicated in visually-guided navigation, as well as the occipital place area (OPA) site. While participants are shown simple visual stimuli of places (e.g., bedrooms, kitchens, and living rooms) they are asked to perform simple computer-based tasks (e.g., imagine they are walking through the room, and respond via button press whether they can leave through a door on the left, center, or right wall, as indicated by a continuous path on the floor). Performance is measured in task accuracy (the percentage of tasks performed correctly). A decrease in performance on the visually-guided navigation task only after rTMS is applied to OPA (but not vertex) indicates causal involvement of OPA in visually-guided navigation.
Time Frame: During rTMS of control site and during rTMS of OPA, on Day 1
Measure: Mean (Standard Deviation); unit: percent of task accuracy
Arm/Group | Repetitive Transcranial Magnetic Stimulation (rTMS) During Computer-based Task
Number analyzed (Participants) | 11
percent of task accuracy
  rTMS Control Site | 80.24 (14.62)
  rTMS Occipital Place Area (OPA) | 82.44 (14.42)

2. Primary Outcome: Reaction Time During Visually-guided Navigation Computer-based Task
Description: To assess performance during the visually-guided navigation computer-based task, rTMS is applied to to the control vertex site, which is not implicated in visually-guided navigation, as well as the occipital place area (OPA) site. While participants are shown simple visual stimuli of places (e.g., bedrooms, kitchens, and living rooms) they are asked to perform simple computer-based tasks (e.g., imagine they are walking through the room, and respond via button press whether they can leave through a door on the left, center, or right wall, as indicated by a continuous path on the floor). Performance is measured in the time (in milliseconds) that it takes to complete the task correctly. A decrease in performance on the visually-guided navigation task only after rTMS is applied to OPA (but not vertex) indicates causal involvement of OPA in visually-guided navigation.
Time Frame: During rTMS of control site and during rTMS of OPA, on Day 1
Measure: Mean (Standard Deviation); unit: milliseconds (ms)
Arm/Group | Repetitive Transcranial Magnetic Stimulation (rTMS) During Computer-based Task
Number analyzed (Participants) | 11
milliseconds (ms)
  rTMS Control Site | 644.23 (120.99)
  rTMS Occipital Place Area (OPA) | 660.08 (109.22)

3. Primary Outcome: Accuracy During Visually-guided Navigation Behavioral-based Task
Description: To assess performance during the visually-guided navigation behavior-based task, rTMS is applied to to the control vertex site, which is not implicated in visually-guided navigation, as well as the occipital place area (OPA) site. Participants are asked to complete simple behavioral-based tasks (e.g., actually walk around a small room and search for hidden objects). Performance is measured in task accuracy (the percentage of tasks performed correctly). A decrease in performance on the visually-guided navigation task only after rTMS is applied to OPA (but not vertex) indicates causal involvement of OPA in visually-guided navigation.
Time Frame: During rTMS of control site and during rTMS of OPA, on Day 1
Population: The study was terminated prior to enrolling participants into the behavioral-based task study arm.
Groups:
- Repetitive Transcranial Magnetic Stimulation (rTMS) During Behavioral-based Task: Participants receiving rTMS while they perform behavioral-based tests to examine the causal involvement of OPA in visually-guided navigation.
Arm/Group | Repetitive Transcranial Magnetic Stimulation (rTMS) During Behavioral-based Task
Number analyzed (Participants) | 0

4. Primary Outcome: Reaction Time During Visually-guided Navigation Behavioral-based Task
Description: To assess performance during the visually-guided navigation behavioral-based task, rTMS is applied to to the control vertex site, which is not implicated in visually-guided navigation, as well as the occipital place area (OPA) site. Participants are asked to complete simple behavioral tasks (e.g., actually walk around a small room and search for hidden objects). Performance is measured as the time (in milliseconds) that it takes to complete the task correctly. A decrease in performance on the visually-guided navigation task only after rTMS is applied to OPA (but not vertex) indicates causal involvement of OPA in visually-guided navigation.
Time Frame: During rTMS of control site and during rTMS of OPA, on Day 1
Population: The study was terminated prior to enrolling participants into the behavioral-based task study arm.
Arm/Group | Repetitive Transcranial Magnetic Stimulation (rTMS) During Behavioral-based Task
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected during the single study visit (Day 1).
Arm/Group | Repetitive Transcranial Magnetic Stimulation (rTMS) During Computer-based Task
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-11): https://cdn.clinicaltrials.gov/large-docs/45/NCT04961645/Prot_SAP_000.pdf
  • Informed Consent Form (2024-06-04): https://cdn.clinicaltrials.gov/large-docs/45/NCT04961645/ICF_001.pdf